CLINICAL TRIAL: NCT02291471
Title: An Open, Dose Escalation, Single Dose Study to Assess Tolerance and Pharmacokinetics of T0001 in Healthy Adult Chinese Volunteers
Brief Title: Tolerance and Pharmacokinetics of T0001 in Healthy Adult Chinese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Fudan-Zhangjiang Bio-Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T0001-P1.0
Record Dates: First submitted 2014-11-11; First posted 2014-11-14 (Estimated); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Rheumatic Diseases
MeSH Terms: conditions — Rheumatic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- T0001 (Experimental)
  Interventions: Drug: T0001，10mg; Drug: T0001，20mg; Drug: T0001，35mg; Drug: T0001，50mg; Drug: T0001，65mg; Drug: T0001，75mg

INTERVENTIONS:
Drug: T0001，10mg
Drug: T0001，20mg
Drug: T0001，35mg
Drug: T0001，50mg
Drug: T0001，65mg
Drug: T0001，75mg

SUMMARY:
The purpose of this study to assess the MTD and Pharmacokinetics of T0001 in Healthy Adult Chinese Volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers, able to give written informed consent for participation in the trial;
* Men or women 50% each , aged 18-45 years old;
* Subjects must have physical examination required and prove medical fitness in 7 days before the clinical starts. BMI should be between 19-24, similar BMI among subjects enrolled at the same time;

Exclusion Criteria:

* Acute or chronic infection, or history of active tuberculosis;
* History of diseases of central nervous system, cardiovascular system, kidney, liver ( specified liver function index), digestive system, respiratory system , metabolism system;
* Subjects who use 5 Unit doses tuberculin skin test are positive( 48-72 hour scleroma reading≥5mm);
* Subjects with a history of mental problems;
* Pregnant and lactating women or women who plan to be pregnant in 3 months;
* Occurence of clinical significant abnormal laboratory examination value during the screening;
* Subjects that lack of understanding ,communication or collaboration, and can't comply with the protocols;
* Subjects that the researchers considered to be not appropriate to participate the trial due to other reasons;

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2014-10; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerance Dose | 3 weeks

SECONDARY OUTCOMES:
Adverse events | 3 weeks
pharmacokinetics parameter(Cmax, AUC, t1/2, CL, etc） | Pre-dose，2、4、12、24、36、48、60、72、84、96、120、144、168、216、264、312、384 and 480hours after the start of subcutaneous injection

CONTACTS AND LOCATIONS:
Overall Officials: Wang wei, Study Director — Shanghai Fudan-Zhangjiang Bio-Pharmaceutical Co., Ltd.; Fang Yi, Ph.D, Principal Investigator — Peking University People's Hospital
Locations (1):
- Phase I laboratory of Peking University People's Hospital, Beijing, Beijing Municipality, China